CLINICAL TRIAL: NCT02054351
Title: A First-in-human Dose Escalation and Dose Finding Phase 1 Trial of IMAB027 in Patients With Recurrent Advanced Ovarian Cancer (OVAR)
Brief Title: Phase 1 Trial of IMAB027 in Patients With Recurrent Advanced Ovarian Cancer (OVAR)
Acronym: OVAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ganymed Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GM-IMAB-002-01; 2013-002755-15 (EudraCT Number); 1650-CL-0101 (Other: Astellas Pharma Global Development, Inc.)
Record Dates: First submitted 2014-01-29; First posted 2014-02-04 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Cancer
Keywords: Advanced ovarian cancer; CLDN6 positive
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMAB027 administration (Experimental): Monotherapy - different dose Levels.
  Interventions: Drug: IMAB027

INTERVENTIONS:
Drug: IMAB027 — Stage 1 (Intrapatient dose escalation): The starting dose is set to 1 mg/m2, followed by 10 mg/m2, 30 mg/m2 and 100 mg/m2 Stage 2 (Interpatient dose escalation): 4 dose level 100 mg/m2, 300 mg/m2, 600 mg/m2, 1000 mg/m2 Extension period: 4 dose level 100 mg/m2, 300 mg/m2, 600 mg/m2, 1000 mg/m2
  Other Names: ASP1650

SUMMARY:
Advanced ovarian cancer is a high medical need indication. Cure is not available to these patients and treatment has palliative intent. A proportion of advanced stage ovarian cancer expresses substantial levels of Claudin 6 (CLDN6), a carcino-embryonic transmembrane protein, which is absent from normal adult human tissue. IMAB027 is a monoclonal antibody that binds to CLDN6. Preclinically IMAB027 was shown to inhibit tumor growth and to kill cancer cells by antibody-dependent cellular cytotoxicity and complement-dependent cytotoxicity. This trial is a first-in-human dose escalation and dose finding Phase 1 trial of IMAB027 in patients with recurrent advanced ovarian cancer to assess the safety and tolerability, the pharmacokinetics, the antitumoral activity and the immunogenicity of IMAB027.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Female patients ≥18 years of age, no upper age limit
3. Histologically or cytologically confirmed CLDN6+ ovarian cancer of any histology type including primary peritoneal or fallopian tube tumors (histological documentation of the original primary tumor is required via a pathology report)
4. Performance status ECOG 0-2
5. Patients with measurable, non-measurable, or evaluable disease: Evaluable disease: defined as a confirmed CA-125 ≥2 x ULN, Measurable disease (RECIST 1.1): defined as at least one lesion that can be accurately measured in at least one dimension
6. Availability of a FFPE tumor tissue sample or tumor cell positive paracentesis fluid samples (abdominal or pleural cavity) for the assessment of CLDN6 positivity
7. Life expectancy of >12 weeks
8. Adequate organ function defined as:

   Adequate hematologic function (ANC ≥1000/μl, platelets ≥100.000/μl, hemoglobin ≥9.0 g/dl (can be post transfusion)); Adequate renal function (serum creatinine ≤1.5 mg/dl [114.5 μmol/l] or creatinine clearance rate ≥30 ml/min); Adequate liver function (serum total bilirubin ≤2 x ULN, AST/ALT ≤3 x ULN)
9. Patients of child-bearing potential must have a negative β-HCG urine test within 72 hours before receiving treatment

Exclusion Criteria:

1. Patient is pregnant or breast-feeding
2. Prior allergic reaction or intolerance to a monoclonal antibody (humanized or chimeric)
3. Any prior anti-tumor therapy within 14 days prior to the start of IMAB027 treatment
4. Other concurrent anticancer therapies
5. HIV infection in medical history or active Hepatitis B or C infection requiring treatment
6. History of any one or more of the following cardiovascular conditions within the past 6 months: Myocardial infarction (T-Wave/Non-T-Wave), Unstable angina pectoris Class II, III or IV congestive heart failure as defined by the New York Heart Association (NYHA), History of cerebrovascular accident, pulmonary embolism or untreated deep venous thrombosis (DVT). Patients with recent DVT who have been or are treated with therapeutic anti-coagulant agents (excluding warfarin) for at least 6 weeks are eligible
7. Other investigational agents or devices concurrently or within 14 days before start of IMAB027 treatment
8. Any hemoptysis or bleeding event that is clinically relevant within 2 weeks of first dose of study drug
9. Clinical symptoms of brain metastases or tumor-associated spinal cord compression
10. Need for continuous, systemic immunosuppressive therapy
11. Any other medical condition that would, in the opinion of the Investigator, limit the patient's ability to complete the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-02-06 (Actual); Primary Completion 2015-10-28 (Actual); Study Completion 2015-10-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 24 month
  Safety profile including type, frequency, severity, relationship of adverse events to investigational medicinal product, dose limiting toxicities, maximum tolerated dose

SECONDARY OUTCOMES:
to assess pharmacokinetics | 24 month
  Cmax, AUC, terminal half-life and related pharmacokinetic parameters of IMAB027
to assess antitumoral activity | up to 3 years
  Disease control rates (CR, PR, SD), ratio previous/current remission time intervals and overall survival
to assess immunogenicity | 24 month
  Frequency of anti-IMAB027 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (9):
- Belgium (2):
  - UZ Brussels, Brussels
  - UZ Leuven, Leuven
- Germany (7):
  - Nationales Centrum für Tumorerkrankungen (NCT) Heidelberg, Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitäts-Frauenklinik (UFK) Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Frauenklinik, Ulm, Baden-Wurttemberg
  - Universitätsmedizin Mainz, Mainz, Rhineland-Palatinate
  - Gemeinschaftspraxis Hämatologie-Onkologie, Dresden, Saxony
  - UKSH Kiel, Kiel, Schleswig-Holstein
  - Charité - Universitätsmedizin Berlin, Berlin

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14577&tenant=MT_AST_9011